CLINICAL TRIAL: NCT04429321
Title: UPCC06820 Phase 1 Trial of Nivolumab + Ipilimumab With Immunostimulatory Embolization for Stage 4 Renal Cell Carcinoma With Unresected Primary
Brief Title: Nivolumab + Ipilimumab With Immunostimulatory Embolization for Stage 4 Renal Cell Carcinoma With Unresected Primary
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: failure to accrue
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06820; 843082 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Renal Cell Carcinoma; Renal Cell Carcinoma Stage IV
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ipilimumab +Nivolumab with Embolization (Experimental): Patients initiate ICI therapy with Nivolumab 3 mg/kg + ipilimumab 1/mg/kg IV every 3 weeks x 4 cycles, followed by nivolumab 480mg flat dose IV every four weeks for a total of 6 months of therapy unless stopped for confirmed progression or intolerable toxicities.
  Patients will receive 2 cycles of systemic therapy followed by embolization of their primary tumor or metastatic lesion(s) and continue systemic therapy subsequently.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Device: bland embolization

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3 mg/kg IV every four weeks, first in combination with capecitabine then alone
  Other Names: Opdivo
Drug: Ipilimumab — ipilimumab 1/mg/kg IV every 3 weeks x 4 cycles, in combination with Nivolumab
  Other Names: Yervoy
Device: bland embolization — Lipiodol:ethanol embolization of their primary or target tumor
  Other Names: trans-arterial embolization

SUMMARY:
This single center phase 1 trial will study the combination of nivolumab+ipilimumab with embolization in participants with renal cell carcinoma. The study will evaluate the safety of embolotherapy in patients with metastatic RCC receiving nivolumab+ipilimumab. The hypothesis is that the number of serious adverse events will be no greater than the number of serious adverse events for both therapies combined.

DETAILED DESCRIPTION:
Previously untreated subjects with stage 4 RCC and unresected primary tumor or metastasis amenable to embolization will undergo two cycles of combination immune checkpoint inhibition (ICI) therapy, embolization of the target tumor, then resume ICI therapy. Study ends with safety and efficacy assessment at 6 months. Correlative blood and tissue specimens will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic renal cell carcinoma with unresected primary tumor or with metastasis amenable to embolization.
2. No prior immune checkpoint therapy
3. Primary tumor or metastasis amenable to percutaneous embolization per review by the treating interventional oncologist

   · Patent feeding artery to tumor > 2 mm diameter without macroscopic arteriovenous fistula/shunt
4. Additional metastatic site > 1 cm assessable for response by RECIST 1.1
5. Adequate organ function by screening laboratory studies within 30 days of embolization

   * platelets > 50K, correctable by transfusion
   * INR < 1.5, correctable by transfusion
   * creatinine < 2.0
6. ECOG performance status 0-2
7. Age ≥ 18 years
8. Have signed the current approved informed consent form and be willing and able to comply with this protocol
9. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of study drug
10. Women of childbearing potential must have a negative serum or urine pregnancy test
11. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose

Exclusion Criteria:

1. Untreated CNS metastasis
2. Autoimmune disorder; subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment
3. Immunodeficiency syndrome
4. Glucocorticoid (> 10 mg daily prednisone equivalents) or immunosuppressant therapy
5. Active infection requiring systemic therapy
6. Any other medical or personal condition that, in the opinion of the site investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical trial.
7. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
8. Contrast allergy not mitigated by usual prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of serious adverse events | Serious adverse events will be recorded from time of informed to consent to 100 days after the end of study intervention
  SAE rate following embolization in patients

SECONDARY OUTCOMES:
Objective response rate | Measured from baseline to 6 months post initiation
  Objective response rate by RECIST 1.1
Characterization of immune cells | From baseline to 12 weeks post initiation of therapy
  Characterization of tumor-infiltrating leukocytes in primary and metastatic lesions before and after embolotherapy
PD-L1 | From baseline to 12 weeks post initiation of therapy
  Percentage of PD-L1 stain positivity in the primary tumor biopsy of participants

CONTACTS AND LOCATIONS:
Overall Officials: Michale Soulen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] Zielinski H, Szmigielski S, Petrovich Z. Comparison of preoperative embolization followed by radical nephrectomy with radical nephrectomy alone for renal cell carcinoma. Am J Clin Oncol. 2000 Feb;23(1):6-12. doi: 10.1097/00000421-200002000-00002. PMID 10683065
- [Background] Swanson DA, Wallace S. Surgery of metastatic renal cell carcinoma and use of renal infarction. Semin Surg Oncol. 1988;4(2):124-8. PMID 3293153
- [Background] Sabel MS. Cryo-immunology: a review of the literature and proposed mechanisms for stimulatory versus suppressive immune responses. Cryobiology. 2009 Feb;58(1):1-11. doi: 10.1016/j.cryobiol.2008.10.126. Epub 2008 Oct 17. PMID 19007768
- [Background] den Brok MH, Sutmuller RP, Nierkens S, Bennink EJ, Frielink C, Toonen LW, Boerman OC, Figdor CG, Ruers TJ, Adema GJ. Efficient loading of dendritic cells following cryo and radiofrequency ablation in combination with immune modulation induces anti-tumour immunity. Br J Cancer. 2006 Oct 9;95(7):896-905. doi: 10.1038/sj.bjc.6603341. Epub 2006 Sep 5. PMID 16953240
- [Background] Mehta A, Oklu R, Sheth RA. Thermal Ablative Therapies and Immune Checkpoint Modulation: Can Locoregional Approaches Effect a Systemic Response? Gastroenterol Res Pract. 2016;2016:9251375. doi: 10.1155/2016/9251375. Epub 2016 Mar 8. PMID 27051417
- [Background] Kato T, Iwasaki T, Uemura M, Nagahara A, Higashihara H, Osuga K, Ikeda Y, Kiyotani K, Park JH, Nonomura N, Nakamura Y. Characterization of the cryoablation-induced immune response in kidney cancer patients. Oncoimmunology. 2017 May 16;6(7):e1326441. doi: 10.1080/2162402X.2017.1326441. eCollection 2017. PMID 28811963